CLINICAL TRIAL: NCT04075760
Title: EUS-guided Combined Therapy of Coiling and 2-octyl-cyanoacrylate Injection With Beta Blocker Therapy Versus Beta Blocker Alone for the Primary Prophylaxis of GOV II and IGV I
Brief Title: EUS-guided Combined Therapy Versus Beta Blocker Therapy in Primary Prophylaxis o GOV II and IGV I
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EUS-PP-GV
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Gastric Varix; Cirrhosis; GastroIntestinal Bleeding
MeSH Terms: conditions — Esophageal and Gastric Varices; Fibrosis; Gastrointestinal Hemorrhage | interventions — Adrenergic beta-Antagonists

STUDY DESIGN:
Intervention Model Description: Randomized control trial, parallel location , 1:1 allocation
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Endoscopic performing EUS evaluation on follow-up will be masked to initial patient allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-guided combined therapy (Experimental): Patients with endoscopic and EUS documented GOV II and IGV I will be included. Procedure will be performed under general anesthesia using a linear array therapeuthic echoendoscope, coils and cyanoacrylate will be injected within the feeder vessel under EUS and fluroscopic guidance.
  Interventions: Procedure: Coils + Cyanoacrylate Group + beta-blocker
- Beta Blocker (Propranolol) (Placebo Comparator): o Beta-blocker (propranolol) will be started at dose of 20 mg twice daily. The principle of incremental dosing was used to achieve the target heart rate for propranolol. The dose will be increased every alternate day to achieve a target heart rate of 55/min or to the maximal dose to 360 mg/day if the medication was well tolerated and the systolic blood pressure was > 90 mm Hg. On the occurrence of intolerable adverse effects, systolic blood pressure < 90 mm Hg or pulse rate < 55/min, the dose of the medication was decreased step-wise, and eventually stopped if these adverse events persisted. Reintroduction of the medication will be attempted if cessation of the medication did not result in improvement of the reported side-effect.
  Interventions: Drug: beta blocker therapy

INTERVENTIONS:
Procedure: Coils + Cyanoacrylate Group + beta-blocker — EUS-combined coiling and cyanoacrylate injection into the feeder vessel of GOV II and IGV I
  Patients with Gastric Varices GOV II or IGV I that have never bleed and are of high-risk GV according to Baveno VI consensus will be prophylactically obliterated via the EUS-guided coiling and cyanoacrylate injection. Patients will also be on beta-blocker therapy as indicated in the other group.
  Arms: EUS-guided combined therapy
Drug: beta blocker therapy — A beta-blocker (propranolol) was started at a dose of 20 mg twice daily. The principle of incremental dosing was used to achieve the target heart rate for propranolol. The dose was increased every alternate day to achieve a target heart rate of 55/min or to the maximal dose to 360 mg/day if the medication was well tolerated and the systolic blood pressure was > 90 mm Hg. On the occurrence of intolerable adverse effects, systolic blood pressure < 90 mm Hg or pulse rate < 55/min, the dose of the medication was decreased step-wise, and eventually stopped if these adverse events persisted. Reintroduction of the medication was attempted if cessation of the medication did not result in improvement of the reported side-effect.
  Arms: Beta Blocker (Propranolol)

SUMMARY:
The EUS-guided combined therapy of coilingand 2-octyl-cyanoacrylate in patients with gastric varices reduced rebleeding and need for reintervention in comparison to EUS-guided coiling alone.The purpose of this study is to determine the efficacy of the primary prophylaxis of GOV II and IGV I with the EUS combined therapy versus beta blocker therapy in patients GOV II and IGV that have never bleed.

DETAILED DESCRIPTION:
Gastric variceal bleeding is a severe condition associated with a high mortality. Bleeding from varices bleeding will be defined as the occurrence of hematemesis and/or melena requiring >2 U of blood or a decrease of 2 gm/dl of hemoglobin if no blood transfusion is given, with the confirmed endocopic visualization of GOV II and IGV I.

The beta blocker therapy is an effective method for the prevention of the first esophageal variceal bleeding; however, the efficacy in preventing first gastric variceal bleeding is controversial.

The investigators aimed to compare the efficacy in preventing the first gastric variceal bleeding in patients with documented GOV II and IGV I.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* Writeen informed consent provided.
* Proven GV (GOV II or IGV I) on esophagogastroduodenoscopy and EUS.
* Gastric varices with high-risk of bleeding (large diameter, high MELD score, presence of portal hypertensive gastropathy)
* Patient preference for EUS-guided therapy.

Exclusion Criteria:

* Under 18 years old.
* Refuse to sign written informed consent.
* Pregnancy or nursing.
* Previous treatment of gastric varices.
* Non-cirrhotic portal hypertension
* Concurrent hepato-renal syndrome and/or multi-organ failure.
* Proven malignancy including hepatocellular carcinoma
* Platelet count less than 50,000/ml or International Normalized Rate (INR) >2.
* Severe ascites that increases the distance between gastric or duodenal and gallbladder walls.
* Esophageal stricture.
* Uncontrolled coagulopathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Bleeding rate secondary to gastric varices | 12 months
  Number of patients with melena or hematemesis accompanied by Hemoglobin drop > 2g/dL
Mortality secondary to gastrointestinal bleeding | 12 months
  mortality rate

SECONDARY OUTCOMES:
Number of reinterventions | 12 months
  number of endoscopic or endoscopic ultrasound procedures requiered for the management of gastri varices

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, M.D., Principal Investigator — Instituto Ecuatoriano de Enfermedades Digestivas
Locations (1):
- Instituto Ecuatoriano de Enfermedades Digestivas, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mishra SR, Sharma BC, Kumar A, Sarin SK. Primary prophylaxis of gastric variceal bleeding comparing cyanoacrylate injection and beta-blockers: a randomized controlled trial. J Hepatol. 2011 Jun;54(6):1161-7. doi: 10.1016/j.jhep.2010.09.031. Epub 2010 Nov 5. PMID 21145834